CLINICAL TRIAL: NCT07148310
Title: Proof-of-Concept Case-Control Study for Hepatocellular Carcinoma Identification Using Delta-HLD Technology (HIDE)
Brief Title: Hepatocellular Carcinoma Identification Using Delta-HLD
Acronym: HIDE
Status: Recruiting | Type: Observational
Sponsor: Epiliquid Holding, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HCC-CPOC; RENIS IS004112 (Other: Epiliquid Holding, Inc)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma; Epigenetics; Liquid Biopsy; cfDNA; Biomarker; Methylation; PCR
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma (cfDNA) samples from whole blood. Hepatocellular carcinoma and cirrhotic liver tissue samples (formalin-fixed and/or fresh-frozen). All samples used for biomarker analysis via delta-HLD
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC-cases: Patients with histologically confirmed hepatocellular carcinoma
- Controls: Patients with liver cirrhosis without evidence of HCC

SUMMARY:
HIDE (Hepatocellular Carcinoma Identification via Delta-HLD) is a proof-of-concept case-control study designed to evaluate the performance of delta-HLD, Epiliquid's proprietary liquid biopsy technology, in detecting hepatocellular carcinoma (HCC). The study includes both plasma and tissue samples to assess biomarker concordance and evaluate diagnostic sensitivity and specificity using tumor-specific methylation markers detected by PCR.

DETAILED DESCRIPTION:
This observational case-control study aims to validate a set of methylation-based biomarkers for HCC detection using delta-HLD technology, which combines enzymatic pre-treatment and multiplexed PCR detection. Epiliquid's proprietary platform also integrates a bioinformatic system that identifies and ranks tumor-specific methylation biomarkers. The study will enroll two groups: patients with histologically confirmed HCC (cases) and patients with liver cirrhosis without evidence of cancer (controls). Liver tissue and blood samples (cfDNA) will be analyzed to assess the sensitivity, specificity, and plasma-tissue concordance of the selected epigenetic signature.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC (cases) or clinically confirmed liver cirrhosis without HCC (controls)
* Willing and able to provide informed consent
* Available paired plasma and liver tissue sample

Exclusion Criteria:

* Other active cancers
* Prior liver transplantation
* Known hereditary cancer syndromes
* Recent chemotherapy or antiviral treatment (<3 months)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be men and women aged 18 years or older, representative of the at-risk population for hepatocellular carcinoma (HCC) in Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of delta-HLD Technology | Within 3 months
  Diagnostic performance of delta-HLD-detected methylation biomarkers in plasma and tissue, using clinical diagnosis of HCC (confirmed by histopathology) as the reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Epiliquid, Mendoza, Argentina

IPD SHARING:
Plan to Share IPD: Undecided